CLINICAL TRIAL: NCT03416751
Title: Fecal Microbial Transplant for Alcohol Misuse in Cirrhosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: OpenBiome (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BAJAJ0021A
Record Dates: First submitted 2018-01-11; First posted 2018-01-31 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Cirrhosis; Alcohol Abuse
MeSH Terms: conditions — Fibrosis; Alcoholism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Fecal Microbial transplantation (Experimental): Patients will get one-dose of 90ml of FMT enema on day 1 that has been received from OpenBiome using a rational donor
  Interventions: Biological: Fecal Microbial Transplant
- Placebo (Placebo Comparator): Patients will get one-dose of 90ml of saline enema on day 1
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Fecal Microbial Transplant — Fecal transplant from a donor in the OpenBiome Registry
  Arms: Fecal Microbial transplantation
Other: Placebo — Placebo enemas
  Arms: Placebo

SUMMARY:
There is an epidemic of alcohol use disorder in the US. Alcoholism is an epidemic that spans all ages and socio-economic strata, which has a major impact on healthcare expenditure. Alcohol-associated liver disease can take the form of mild fatty liver, chronic liver disease including cirrhosis and a very acute active form known as alcoholic hepatitis. However, most patients with alcohol abuse issues with cirrhosis do not develop alcoholic hepatitis and are not willing to quit drinking. These patients are neither liver transplant candidates due to their drinking nor have any recourse to therapies directed towards the liver as is the case with alcoholic hepatitis. This is very large proportion of cirrhotic patients who do not have many therapeutic options.

Prior studies have demonstrated that these patients have an altered gut-liver axis which is exacerbated by dysbiosis and a higher production of potentially toxic secondary bile acids. These secondary bile acids in turn have the potential to worsen the already impaired gut barrier in these patients, creating a vicious cycle of inflammation and further liver injury that is led by the altered microbial composition. A gut-based strategy that has the capability of "resetting" this dysbiosis could help in the amelioration of this inflammatory load and improve the prognosis of these patients.

DETAILED DESCRIPTION:
Randomized, single-blind, placebo-controlled safety, tolerability study with exploratory endpoints and pathophysiological evaluation of the FMT

Two groups of outpatients with cirrhosis will be randomized using random sequence generator into no-treatment and FMT groups.

Once patients are randomized 1:1 into group 1 (FMT) and group 2 (Placebo), both will be followed over 31 days and will include a 6 month visit to collect samples, perform questionnaires and to assess SAEs.

There is an epidemic of alcohol use disorder in the US. Alcoholism is an epidemic that spans all ages and socio-economic strata, which has a major impact on healthcare expenditure. Alcohol-associated liver disease can take the form of mild fatty liver, chronic liver disease including cirrhosis and a very acute active form known as alcoholic hepatitis. However, most patients with alcohol abuse issues with cirrhosis do not develop alcoholic hepatitis and are not willing to quit drinking. These patients are neither liver transplant candidates due to their drinking nor have any recourse to therapies directed towards the liver as is the case with alcoholic hepatitis. This is very large proportion of cirrhotic patients who do not have many therapeutic options.

Prior studies have demonstrated that these patients have an altered gut-liver axis which is exacerbated by dysbiosis and a higher production of potentially toxic secondary bile acids. These secondary bile acids in turn have the potential to worsen the already impaired gut barrier in these patients, creating a vicious cycle of inflammation and further liver injury that is led by the altered microbial composition. The investigators believe that a gut-based strategy that has the capability of "resetting" this dysbiosis can help in the amelioration of this inflammatory load and improve the prognosis of these patients.

ELIGIBILITY:
Inclusion Criteria:

A. Cirrhosis diagnosed by any of the following in a patient with chronic liver disease:

1. Liver Biopsy
2. Radiologic evidence of varices, cirrhosis or portal hypertension
3. Laboratory evidence of platelet count <100,000 or AST/ALT ratio>1
4. Endoscopic evidence of varices or portal gastropathy
5. Fibroscan B. Age between 21 and 75 C. Able to give written, informed consent (demonstrated by mini-mental status exam>25 at the time of consenting) D. Subject must have alcohol as a cause of cirrhosis

i. Continued sustained drinking pattern with AUDIT score ≥8 in the last month and fulfilling DSM-V criteria for alcohol misuse ii. Unable or unwilling to get mental health attention to quit alcohol (at least 3-months period of referrals to Substance abuse programs or other alcohol treatment approaches) iii. Adult companion who can accompany patient and provide insight into alcohol drinking patterns

Exclusion Criteria:

A. MELD score >17 B. Child Class C C. WBC count <1000 cells/mm3 D. Platelet count<50,000/mm3 E. TIPS in place for less than a month F. HE episode within a month prior to the study G. Currently on absorbable antibiotics H. Infection at the time of the FMT (diagnosed by blood culture positivity, urinalysis, paracentesis as needed) I. Patients who are aged >75 years J. Patients who are pregnant or nursing (will be checked using a urine pregnancy test) K. Patients who are incarcerated L. Patients who are incapable of giving their own informed consent

M. Patients who are immuno-compromised due to the following reasons:

1. HIV infection (any CD4 count)
2. Inherited/primary immune disorders
3. Current or recent (<3 months) treatment with anti-neoplastic agent
4. Current or recent (<3 months) treatment with any immunosuppressant medications [including but not limited to monoclonal antibodies to B and T cells, anti-TNF agents, glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine), calcineurin inhibitors (tacrolimus, cyclosporine), mycophenolate mofetil]. Subjects who are otherwise immunocompetent and have discontinued any immunosuppressant medications 3 or more months prior to enrollment may be eligible to enroll.

N. Patients with a history of severe (anaphylactic) food allergy O. Patients who have previously undergone FMT P. Patients on renal replacement therapy Q. Patients who are unwilling or unable to hold the enemas R. Patients with untreated, in-situ colorectal cancer S. Patients with a history of chronic intrinsic GI diseases such as inflammatory bowel disease (ulcerative colitis, Crohn's disease or microscopic colitis), eosinophilic gastroenteritis, celiac disease or irritable bowel syndrome T. Major gastro-intestinal or intra-abdominal surgery in the last three months U. Unable to comply with protocol requirements V. Patients who are American Society of Anesthesiologists (ASA) Physical Status classification IV and V W. Patients with acute illness or fever on the day of planned FMT will be excluded with the option of including that subject at a future date X. Any conditions for which, in opinion of MD, the treatment may pose a health risk Y. Grade 2-4 or complicated hemorrhoids

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-04-10 (Actual); Study Completion 2020-04-10 (Actual)

PRIMARY OUTCOMES:
Proportion of participants with a related serious adverse event | 15 days
  Related SAE to FMT
Proportion of participants with newly acquired transmissible infectious diseases | 15 days
  Related transmissible infectious disease to FMT
Proportion of participants with a related adverse event | 15 days
  Related adverse event that does not meet the criteria for a serious adverse event

SECONDARY OUTCOMES:
Proportion of participants with a related serious adverse event | 30 days and 6 months
  Related SAE to FMT
Proportion of participants with a related adverse event | 30 days and 6 months
  Related adverse event that does not meet the criteria for a serious adverse event
Proportion of participants with newly acquired transmissible infectious diseases | 30 days and 6 months
  Related transmissible infectious disease to FMT
Composition of microbial change | day 15 post-intervention
  UNIFRAC and LEFSe pre vs post FMT on stool microbiota compared to baseline and to placebo
AUDIT questionnaire | day 15 post-intervention
  defining changes in alcohol abuse severity compared to baseline and to placebo
Alcohol craving questionnaire | day 15 post-intervention
  defining changes in the cravings for alcohol compared to baseline and to placebo
Systemic inflammation changes | day 15 post-intervention
  Inflammatory cytokines (IL-6, TNF, IL-1b) compared to baseline and to placebo
Cognition change using PHES | day 15 post-intervention
  Psychometric hepatic encephalopathy score compared to baseline and to placebo
Cognition change using EncephalApp stroop | day 15, 30 and 6 months post-intervention
  EncephalApp stroop compared to baseline and to placebo
Quality of Life using Sickness Impact Profile | day 15 post-intervention
  Sickness Impact Profile compared to baseline and to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Jasmohan S Bajaj, MD, Principal Investigator — Hunter Holmes McGuire VA Medical Center
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided